CLINICAL TRIAL: NCT04442984
Title: FOLFOX6 Versus mFOLFIRINOX as First Line Chemotherapy in Metastatic Gastric or Esophagogastric Junction Adenocarcinoma (Type II-III): Open-label Randomized Phase 2/3 Trial
Brief Title: FOLFOX6 Versus mFOLFIRINOX as First Line Chemotherapy in Metastatic Gastric Cancer or Esophagogastric Junction Adenocarcinoma (Type II-III)
Acronym: IRIGA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Gastric Carcinoma Stage IV; Esophagogastric Junction Adenocarcinoma Stage IV
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFOX6 (Active Comparator): 5FU 400mg/m2 iv bolus d1, 5-FU 2400 mg/m² d1-2, Leucovorin 400 mg d1, Oxaliplatin 85 mg/m² d1, every two weeks (q2w) 9 cycles
  Interventions: Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-FU
- mFOLFIRINOX (Experimental): Irinotecan 180mg/m2 d1, 5FU 250mg/m2 iv bolus d1, 5-FU 2200 mg/m² d1-2, Leucovorin 400 mg d1, Oxaliplatin 85 mg/m² d1, every two weeks (q2w) 9 cycles
  Interventions: Drug: Irinotecan; Drug: Oxaliplatin; Drug: 5-FU; Drug: Leucovorin

INTERVENTIONS:
Drug: Irinotecan — d1 Irinotecan 180mg/m² every two weeks
  Arms: mFOLFIRINOX
Drug: Oxaliplatin — d1 Oxaliplatin 85 mg/m² every two weeks
Drug: 5-FU — d1-2 5-FU 2200 mg/m² every two weeks
  Arms: mFOLFIRINOX
Drug: 5-FU — d1 5-FU 250 mg/m² every two weeks
  Arms: mFOLFIRINOX
Drug: Leucovorin — d1 Leucovorin 400 mg every two weeks
Drug: 5-FU — d1 5-FU 400 mg/m² every two weeks
  Arms: FOLFOX6
Drug: 5-FU — d1-2 5-FU 2400 mg/m² every two weeks
  Arms: FOLFOX6

SUMMARY:
Patients with metastatic adenocarcinoma of the stomach or the esophagogastric junction (II-III type by Siewert) without previous therapy will be treated with one of two chemotherapy combinations . One half of the patients gets 5-Fluorouracil (5-FU), Leucovorin, Oxaliplatin (FOLFOX6), the others 5-Fluorouracil (5-FU), Leucovorin, Oxaliplatin and Irinotecan (mFOLFIRINOX). Main objective of the study is progression free survival.

DETAILED DESCRIPTION:
This parallel, randomized, open-label study 326 patients with metastatic ( adenocarcinoma of the stomach or the esophagogastric junction without previous therapy will be included in this study. After randomization patients receive 9 cycles FOLFOX6 or mFOLFIRINOX.

Stratification factors include ECOG, site of metastasis, age, pathological subtypes.

Efficacy will be evaluated every 3 cycles with RECIST. Toxicity will be assessed with WHO CTC 3.0 every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed locally advanced, recurrent or metastatic adenocarcinoma of the esophagogastric junction (Siewert type II-III) or the stomach
2. no prior palliative chemotherapy or radiation therapy
3. Age 18-70 years (female and male)
4. Eastern Cooperative Oncology Group ≤ 2
5. Neutrophils> 2.000/µl
6. Platelets > 100.000/µl
7. Normal value of Serum Creatinin
8. Albumin level > 29 г/л
9. Aspartate transaminase (AST) or alanine transaminase (ALT) less than 3 times the upper limits of normal (ULN)
10. Total Bilirubin less than 1.5 times the ULN
11. Written informed consent.

Exclusion Criteria:

1. Previous palliative cytostatic chemotherapy
2. Cancer relapse
3. Complicated gastric cancer (perforation, bleeding, sub or decompensated stenosis, dysphagia IV)
4. Diarrhea ≥ 2 according to the criteria of Common Terminology Criteria for Adverse Events (CTCAE) version 4.1;
5. Hypersensitivity against 5- Fluorouracil, Leucovorin, Oxaliplatin, irinotecan
6. Existence of contraindications against 5- Fluorouracil, Leucovorin, Oxaliplatin, Irinotecan or Docetaxel
7. Active coronary heart disease, Cardiomyopathy or cardiac insufficiency stage III-IV according to New York Heart Association (NYHA)
8. Severe non-surgical accompanying disease or acute infection (uncontrolled arterial hypertension, diabetes mellitus, stroke less than 6 months old, mental disorders, other tumors and others)
9. Malignant secondary disease, dated back < 5 years (exception: In-situ-carcinoma of the cervix uteri, adequately treated skin basal cell carcinoma)
10. Peripheral polyneuropathy > Grad II
11. Liver dysfunction (AST)/ALT>3,0xULN, ALT>3xULN, Bilirubin>1,5xULN) Serum Creatinin >1,0xULN
12. Chronic inflammable gastro-intestinal disease
13. Inclusion in another clinical trial
14. Pregnancy or lactation
15. Hepatitis B or C in the active stage
16. Human immunodeficiency virus(HIV) infected
17. Serious concomitant somatic and mental illnesses / deviations or territorial causes that may prevent the patient from participating in the protocol and observing the protocol schedule
18. Foreigners or persons with limited legal status

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 326 (Estimated)
Dates: Start 2019-11-03 (Actual); Primary Completion 2021-11-03 (Estimated); Study Completion 2024-11-03 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | 36 months
  PFS is defined as the time from the date of randomization to the date of the first documentation of progressive disease or date of death, whichever occurs first. For target lesions (TL), PD was defined as at least a 20 percent (%) increase in the sum of the longest diameter (SLD) of TLs, taking as a reference the smallest SLD recorded since the treatment started, or the appearance of one or more lesions. For non-target lesions (NTL), PD was defined as an unequivocal progression of existing NTLs. Participants were censored at the last date of tumor measurement, the last date in the study drug log, or the date of last follow-up.

SECONDARY OUTCOMES:
Overall Survival (OS) | 60 months
  OS is defined as the time from the date of randomization to the date of death due to any cause. Participants were censored at the last date of tumor measurement, the last date in the study drug log or the date of last follow-up
Percentage of Participants With Confirmed Complete Response (CR) or Partial Response (PR) Determined by Response Evaluation Criteria in Solid Tumors (RECIST) | 12 months
Duration of Response | 12 months
Treatment associated toxicities | 12 months
  WHO CTC 3.0

CONTACTS AND LOCATIONS:
Locations (1):
- Blokhin's Russian Cancer Research Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No